CLINICAL TRIAL: NCT01135628
Title: Hyperproteic and Fiber-rich Diet Plus Probiotics (Lactobacillus Reuteri) and Nitazoxanide in the Treatment of Minimal Hepatic Encephalopathy.
Brief Title: Hyperproteic Diet Plus Lactobacillus Reuteri and Nitazoxanide in Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D. M.Sc, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAS-83-09/10-1
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Hepatic Cirrhosis; Minimal Hepatic Encephalopathy
Keywords: Hepatic cirrhosis; Minimal hepatic encephalopathy; Hyperproteic and fiber-rich diet; Lactobacillus reuteri; Psychometric Hepatic Encephalopathy Score (PHES); Critical Flicker Frequency (CFF)
MeSH Terms: conditions — Liver Cirrhosis | interventions — Probiotics; nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MHE and diet plus lactobacillus reuteri (Active Comparator): Patients with minimal hepatic encephalopathy managed with diet consisting in hyperproteic and fiber-rich foods and lactobacillus reuteri.
  Interventions: Other: Auxiliary Treatment; Dietary Supplement: Hyperproteic and fiber-rich diet
- MHE and diet (Active Comparator): Patients with minimal hepatic encephalopathy managed with diet consisting in hyperproteic and fiber-rich foods.
  Interventions: Dietary Supplement: Hyperproteic and fiber-rich diet
- MHE and diet plus nitazoxanide (Active Comparator): Patients with minimal hepatic encephalopathy managed with diet consisting in hyperproteic and fiber-rich foods and nitazoxanide.
  Interventions: Dietary Supplement: Hyperproteic and fiber-rich diet; Drug: Nitazoxanide

INTERVENTIONS:
Other: Auxiliary Treatment — Lactobacillus reuteri, 1 tablet bid, each of 100,000,000 FCU for 6 months
  Other Names: Biogaia; Probiotics
  Arms: MHE and diet plus lactobacillus reuteri
Dietary Supplement: Hyperproteic and fiber-rich diet — Hyperproteic diet consisting in 1.5 gr/kg of protein per day Fiber-rich diet
Drug: Nitazoxanide — Nitazoxanide tablets 400 mg, bid, orally for 6 months
  Arms: MHE and diet plus nitazoxanide

SUMMARY:
Hepatic encephalopathy is a serious complication of cirrhosis which relays under the burden of diseases with therapeutical difficulties for its given morbidity and mortality and the high recurrence it poses. Its treatment remains a challenge for most of the cases. Even more, minimal hepatic encephalopathy is an entity that has an additional morbidity for it being a subclinical entity. As so, the investigators propose an auxiliary treatment for the management of such patients with minimal hepatic encephalopathy, using a specific diet consisting on hyperproteic and fibre-rich foods along with two independent interventions, whether a probiotic, lactobacillus reuteri, or a drug, nitozoxanide, so to diminish the rate of progression to any clinical stage of hepatic encephalopathy and to revert minimal hepatic encephalopathy itself to none hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic Cirrhosis
* Minimal hepatic Encephalopathy

Exclusion Criteria:

* Personal history of surgery in the last 4 weeks
* Use of neuropsychiatric drugs
* Neuropsychiatric disorders (Schizophrenia, bipolar disorder, major depression, dementia and Attention-deficit hyperactivity disorder)
* Thyroid disorders without replacement therapy
* Hepatic or renal transplant
* Alcoholism with active ingest of alcohol in the last 6 months
* Pregnancy
* Labour turn-overs
* Spontaneous bacterial Peritonitis
* Personal history of hepatocellular carcinoma
* Placement of transjugular intrahepatic portosystemic shunt
* Use of a probiotic in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reverse minimal hepatic encephalopathy | 3 months
  Reverse minimal hepatic encephalopathy to none evidence of hepatic encephalopathy
Reverse minimal hepatic encephalopathy | 6 months
  Reverse minimal hepatic encephalopathy to none evidence of clinical hepatic encephalopathy

SECONDARY OUTCOMES:
Prevention of progression | 3 months
  Prevention of progression from minimal hepatic encephalopathy to any clinical stage of West Haven score of hepatic encephalopathy.
Prevention of progression | 6 months
  Prevention of progression from minimal hepatic encephalopathy to any clinical stage of West Haven score of hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre-Delgadillo, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas de Nutricion
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico